CLINICAL TRIAL: NCT05828940
Title: The Effect of Losartan on Emotion Regulation
Brief Title: Losartan and Memory
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oxford (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: R58494/RE003
Record Dates: First submitted 2023-04-12; First posted 2023-04-25 (Actual); Last update posted 2023-04-27 (Actual); Status verified 2023-04

CONDITIONS: PTSD
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — Losartan

STUDY DESIGN:
Intervention Model Description: randomised double-blind
Who Masked: Participant, Investigator
Masking Description: double-blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- placebo (Placebo Comparator): microcellulose
  Interventions: Drug: Placebo
- losartan (Experimental): 50mg losartan (Cozaar)
  Interventions: Drug: Losartan Potassium

INTERVENTIONS:
Drug: Losartan Potassium — oral tablet, over-encapsulated
  Arms: losartan
Drug: Placebo — oral tablet, over-encapuslated
  Arms: placebo

SUMMARY:
This study investigates the effect of a single dose of 50mg losartan vs placebo on BOLD signal during memory encoding.

DETAILED DESCRIPTION:
The commonly prescribed antihypertensive drug losartan targets the renin-angiotensin system - a hormone system regulating blood pressure - by acting as an angiotensin receptor antagonist. The drug prevents a docking of the protein angiotensin IV to AT1 receptors, which leads to a dilation if vessels and a reduction in blood pressure. However, the increase in free angiotensin IV has also been associated with an increase in synaptic plasticity, the cellular mechanism involved in learning and memory. As such, losartan appears to have cognition-enhancing properties, in a way that a single dose of 50mg improves prospective memory in healthy humans . However, preliminary pre-clinical results also suggest that a single injection of the drug improves fear extinction in rodents, which is the equivalent to human cognitive-behavioural therapy for anxiety disorders . Furthermore, compared to other antihypertensive drugs, regular losartan treatment appears to prevent the development of post-traumatic stress disorder following trauma exposition . Such results suggest that the renin-angiotensin system may play a key role in the prevention of anxiety.

In this study, we investigate the effect kof probing the renin-angiotensin system on memory encoding, which has previously been shown to be impaired in PTSD. In a double-blind, randomised between-groups design, 40 healthy volunteers with moderate to high levels of trait anxiety are randomised to a group receiving a single dose of losartan (50mg) versus placebo. When peak plasma levels are reached, participants work on a battery of behavioural and neural measures of emotional information processing. These tasks will include an fMRI task where participants will see images of animals and landscapes on the screen and categorise these accordingly, to be tested for memory for these images in a later task.

The results from this study will help us understand how the renin-angiotensin system affects memory formation, and they will help us establish a battery of tasks that sensitively respond to such manipulations. Such information will ultimately lead to the development of losartan and similar agents for the more effective and more compact treatment of anxiety disorders.

ELIGIBILITY:
Inclusion Criteria:

* willing and able to provide informed consent
* male or Female, aged 18-50 years
* body mass index (BMI) of 18-30 kg/m2
* non- or light-smoker (< 5 cigarettes a day)
* STAIT score of at least 40

Exclusion Criteria:

* Female participant who is pregnant or breast-feeding
* CNS-active medication during the last 6 weeks
* Current blood pressure or other heart medication (especially aliskiren or beta blockers)
* Diagnosis of intravascular fluid depletion or dehydration
* Past or present DSM-IV axis-I diagnosis or suspected diagnosis (from SCID results at screening)
* Alcohol or substance abuse
* First-degree family member with a history of a severe psychiatric disease
* Impaired liver or kidney function
* Lifetime history of epilepsy or other neurological disease, systemic infection, or clinically significant hepatic, cardiac, obstructive respiratory, renal, cerebrovascular, metabolic, endocrine or pulmonary disease or disorder which, in the opinion of the investigator, may either put the participants at risk because of participation in the study, or may influence the result of the study, or the participant's ability to participate in the study.
* High or moderate risk of coronavirus, based on the NHS checklist for coronavirus vulnerability https://www.nhs.uk/conditions/coronavirus-covid-19/people-at-higher-risk/whos-at-higher-risk-from-coronavirus/
* Contraindication to MRI (e.g. metal implant)
* Insufficient English skills
* participated in another study involving CNS-active medication during the last 6 weeks Participants will also not be able to take part if they are left-handed, due to the research MRI aspect of the study relying on group means.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 41 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2022-03-31 (Actual); Study Completion 2022-03-31 (Actual)

PRIMARY OUTCOMES:
BOLD activation in hippocampus during new>familiar contrast | one hour after capsule intake

SECONDARY OUTCOMES:
BOLD activation in other brain areas | one hour after capsule intake
pattern similarity | one hour after capsule intake

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Reinecke, PhD, Principal Investigator — Unoversity of Oxford
Locations (1):
- Department of Psychiatry, University of Oxford, Oxford, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Data may be shared upon reasonable request, and within the conditions of our ethics approval.